CLINICAL TRIAL: NCT02213731
Title: Cryoballoon Ablation for Early Persistent Atrial Fibrillation
Brief Title: Cryoballoon Ablation for Early Persistent Atrial Fibrillation (Cryo4 Persistent AF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cryo4 Persistent AF
Record Dates: First submitted 2014-07-31; First posted 2014-08-11 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Persistent Atrial Fibrillation; Cryoablation; Cryoballoon; Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoballoon ablation (Other): Subjects will wear holter monitors at baseline, 6 months and 12 months
  Interventions: Other: Holter monitoring

INTERVENTIONS:
Other: Holter monitoring — Subjects will wear holter monitors at baseline, 6 months and 12 months.

SUMMARY:
The purpose of this clinical study is to assess the single procedure outcomes of using cryoballoon ablation without additional empirical lesions and/or complex fractionated electrogram (CFE) ablations for patients with early persistent atrial fibrillation (<1 year from first diagnosis of persistent AF).

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented symptomatic persistent AF refractory or intolerant to at least 1 class I or III antiarrhythmic medication. Persistent AF defined as:

  * Episode lasting longer than 7 days, but less than 1 year documented by consecutive ECG recordings of 100% AF greater than 7 days apart OR
  * Episode requiring electrical or pharmacological cardioversion after 48 hours of AF documented by continuous recording
* Date of first diagnosis of persistent AF within the last 12 months preceding the consent date
* Age between 18 and 75 years
* Willing to comply with study requirements and give informed consent (defined as legally effective, documented confirmation of a subject's (or their legally authorized representative or guardian) voluntary agreement to participate in a particular clinical study) to participate in this clinical study

Exclusion Criteria:

* Long-standing persistent AF (has lasted for ≥1 year)
* Current diagnosis of paroxysmal AF
* Anteroposterior LA diameter > 5.0 cm by TTE
* Current intracardiac thrombus
* Presence of one or more pulmonary vein stents
* Presence of any pre-existing pulmonary vein stenosis
* Primary pulmonary hypertension
* NYHA class IV congestive heart failure and/or documented left ventricular ejection fraction (LVEF) < 40% measure by acceptable cardiac testing (e.g. TTE)
* Hypertrophic cardiomyopathy
* Previous LA ablation or surgery
* Unstable angina
* Presence of any cardiac valve prosthesis
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* Any cardiac surgery, myocardial infarction, PCI / PTCA or coronary artery stenting which occurred during the 3 month interval preceding the consent date
* Any cerebral ischemic event (strokes or TIAs) which occurred during the 6 month interval preceding the consent date
* Cryoglobulinemia
* Presence or likely implant of a permanent pacemaker, biventricular pacemaker, loop recorder, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) within 12 months
* Uncontrolled hyperthyroidism
* Any woman known to be pregnant or breastfeeding
* Active systemic infection
* Subject is employed by Medtronic or by the department of any of the investigators or is a close relative of any of the investigators
* Life expectancy ≤ 1 year
* Currently enrolled or plans to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent studies is allowed when documented pre-approval is obtained from the Medtronic study manager
* Exclusion criteria as per local laws (for France, this includes, but is not limited to: incompetent adults or patients that are not affiliated to the French social security system)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Single procedure success of cryoballoon ablation on patients with early persistent AF | 12 months
  12 month success will be defined as absence of adjudicated AF/atrial flutter/atrial tachyarrhythmias >/= 30 seconds in duration from the end of the 90 day blanking period of the cryoballoon ablation procedure to at least 12 months after the cryoballoon ablation procedure. Only Arctic Front Advance catheters may be used to achieve the single procedure success and no additional empirical lesions and/or complex fractionated electrogram (CFE) ablations may be made. Additionally, subjects must not require any other intervention for AF following the index procedure. Right atrial flutter ablations and pharmacological and/or electrical cardioversion can be performed within the 90 day blanking period.

SECONDARY OUTCOMES:
Acute procedural success of cryoballoon ablation on patients with early persistent AF | Post-procedure
  Acute procedural success is defined as:
  * Only Arctic Front Advance catheters used to achieve procedure success AND
  * All targeted pulmonary veins were isolated (minimally assessed for entrance block and, where assessable, exit block) AND
  * Sinus rhythm is restored at the end of the ablation procedure (with or without cardioversion)
Success of cryoballoon ablation on patients with early persistent AF (allowing for multiple procedures) | 12 months
  12 month success will be defined as absence of adjudicated AF/atrial flutter/atrial tachyarrhythmias >/= 30 seconds in duration from the end of the 90 day blanking period of the cryoballoon ablation procedure to at least 12 months after the cryoballoon ablation procedure. Only Arctic Front Advance catheters may be used to achieve multiple procedure success and no additional empirical lesions and/or complex fractionated electrogram (CFE) ablations may be made. Additionally, subjects must not require any other intervention for AF. Right atrial flutter ablations and pharmacological and/or electrical cardioversion can be performed within the 90 day blanking period.
Sinus rhythm restoration being followed by chronic prevention of AF recurrence | 12 months
Use of class I and class III antiarrhythmic drugs | 12 months
Changes in quality of life measurements between baseline, 6 months and 12 months after procedure | Baseline, 6 months, 12 months
Adverse events required to be collected during the study | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Serge Boveda, M.D., Principal Investigator — Clinique Pasteur; Pascal Defaye, M.D., Principal Investigator — CHU Michallo, Unité de Rythmologie, Clinique de cardiologie, CHU de Grenoble site Nord - Hôpital Albert Michallon
Locations (14):
- France (5):
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CHU de la Timone, Marseille
  - CHU - Hôpitaux de Rouen, Rouen
  - Clinique Pasteur, Toulouse
- Germany (8):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charite - Universitaetsmedizin, Berlin
  - Krankenhaus Porz am Rhein, Cologne
  - St. Vinzenz-Hospital, Cologne
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Asklepios Klinik St. Georg, Hamburg
  - Klinikum Nürnberg Süd, Nuremberg
  - Uniklinik Ulm, Ulm
- Henry Dunant Hospital Center, Athens, Greece

REFERENCES:
- [Derived] Boveda S, Metzner A, Nguyen DQ, Chun KRJ, Goehl K, Noelker G, Deharo JC, Andrikopoulos G, Dahme T, Lellouche N, Defaye P. Single-Procedure Outcomes and Quality-of-Life Improvement 12 Months Post-Cryoballoon Ablation in Persistent Atrial Fibrillation: Results From the Multicenter CRYO4PERSISTENT AF Trial. JACC Clin Electrophysiol. 2018 Nov;4(11):1440-1447. doi: 10.1016/j.jacep.2018.07.007. Epub 2018 Aug 25. PMID 30466850